CLINICAL TRIAL: NCT04900298
Title: Reducing Intraoperative ESKAPE (Enterococcus, S. Aureus, Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter Spp.) Transmission in the Adult Operating Room Via Use of a Personal Hand Hygiene System Optimized by OR PathTrac
Brief Title: Reducing Intraoperative ESKAPE Transmission Through Use of a Personal Hand Hygiene System
Acronym: ESKAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Georgia-Pacific Consumer Products LP (Unknown); University of Iowa (Other); RDB Informatics (Unknown)
Responsible Party: Principal Investigator, Brandon M Togioka, Principal Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 22966
Record Dates: First submitted 2021-05-12; First posted 2021-05-25 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Surgical Wound Infection; Cross Infection
MeSH Terms: conditions — Surgical Wound Infection; Cross Infection

STUDY DESIGN:
Intervention Model Description: This will be a prospective, single center, unmasked, controlled before and after study. Two patients (case-pair) having surgery in a serial manner in a randomly selected operating room will be evaluated for the detection of pathogenic bacteria. The first twenty patients (10 case-pairs) will be enrolled in the control (standard care) arm followed by 20 patients (10 case-pairs) being enrolled in the intervention (SafeHaven) arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Use of SafeHaven hand hygiene system in the operating room
  Interventions: Device: SafeHaven Automated Hand Hygiene Device
- Control Arm (No Intervention): Standard of care hand hygiene

INTERVENTIONS:
Device: SafeHaven Automated Hand Hygiene Device — Anesthesia providers in the intervention arm will be given a personal hand hygiene device, containing 64% ethyl alcohol, which provides actionable real-time performance feedback. The personalized device will be affixed to the provider's waist and will remain there for use throughout the perioperative period. Performance feedback is given to the anesthesia provider in real time with the number of personal hand hygiene events and an hourly hand hygiene rate, which is displayed on the device. Devices will be handed out to participating providers in the preoperative bay and retrieved in the post-anesthesia care unit upon case completion.
  Arms: Intervention Arm

SUMMARY:
The investigators hypothesize that the use of a personal hand hygiene system (SafeHavenTM) by anesthesia providers in the adult operating room, combined with a novel infectious pathogen tracking system (OR PathTrac) will decrease participant exposure to pathologic bacteria in the adult operating room.

DETAILED DESCRIPTION:
This will be a prospective, single center, unmasked, controlled before and after study.

Intervention Arm: Use of SafeHaven hand hygiene system in the operating room

Control Arm: Standard of care hand hygiene

Operating Room Selection: Two patients (case-pair) having surgery in a serial manner in a randomly selected operating room will be evaluated for detection of pathogenic bacteria. The operating room for investigation will be randomly selected through the following process:

1. All the operating rooms with scheduled surgeries in the South Operating Rooms on a particular day will be entered into a random number generator (example: operating rooms 2, 3, 5, 7).
2. The random generator will sort these operating rooms into a rank list (example: operating rooms 5, 3, 2, 7).
3. The investigators will start at the top of this list and work down until the first operating room meeting all inclusion criteria is found (example: operating room 5 only has one surgery, operating room 3 has pediatric surgery, operating room 2 meets inclusion criteria)
4. This process will be duplicated for each case-pair

The goal of the study is to map transmission of bacteria through the operating room and compare mapping with the SafeHaven Hand Hygiene system to mapping without the SafeHaven Hand Hygiene system. Thus, case-pairs will be randomized to the same assignment. For example, subject 1 and 2 will have surgery in South Operating Room 8 and both will be randomized to the control group. The first 10 case-pairs will be assigned to the control arm and the second 10 case-pairs will be assigned to the intervention arm.

ELIGIBILITY:
Patient Inclusion Criteria:

Patients ≥ 18 years of age having surgery in an adult operating suite at the research center involving the following specialties: orthopedics/spine, orthopedics/total joint, gynecology/oncology, colorectal, open vascular, and open urological, general abdominal, acute care, cardiothoracic, and plastic/breast.

Patient Exclusion Criteria:

* Patients with a known infection at the time of surgery.
* Prisoners
* Pregnant Women
* Patients lacking capacity to consent
* Patients with an allergy to a component of hand hygiene solution, such as ethyl alcohol
* Refusal of consent

Anesthesia Provider Inclusion Criteria:

• Faculty physicians, resident physicians, or certified registered nurse anesthetists that provide care for adults having surgery at the research center.

Anesthesia Provider Exclusion Criteria:

* Refusal of consent
* Open sores of the hands
* Known skin infection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of ESKAPE (Enterococcus, S. Aureus, Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter spp.) reservoirs identified using microbial culture collection kits | Perioperative Time, typically less than 12 hours
  The following reservoirs will be cultured at case start (anesthesia machine adjustable pressure limiting valve, patient nare, patient axilla, patient groin, anesthesia provider dominant hand, primary assigned anesthesia assistant) and at case end (anesthesia machine adjustable pressure limiting valve, patient nare, patient axilla, patient groin, anesthesia provider dominant hand, primary assigned anesthesia assistant, and internal lumen of intravenous tubing stopcock) within the operating room suite using a sterile collection kit.

SECONDARY OUTCOMES:
Number of ESKAPE (Enterococcus, S. Aureus, Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter spp.) transmission events using OR PathTrac Software. | 30 days following surgery
  OR Path Trac software algorithms will map how ESKAPE pathogens are transmitted from an initially identified reservoir to a new location within the perioperative environment.
Quantitate the reduction in ESKAPE (Enterococcus, S. Aureus, Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter spp.) transmission events | 30 days following surgery
  Compare the reduction in ESKAPE transmission events for patients who receive standard of care versus patients who have anesthesia providers that use the SafeHaven personal hand hygiene device

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Togioka, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.